CLINICAL TRIAL: NCT03048383
Title: Randomized, Single-blind Comparison of Three Commercially Available Botulinum Neuromodulators in the Management of Facial Synkinesis
Brief Title: Comparison of Three Botulinum Neuromodulators for Management of Facial Synkinesis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Preston Ward, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 56158
Record Dates: First submitted 2017-02-02; First posted 2017-02-09 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-06

CONDITIONS: Facial Nerve Injuries; Facial Paresis Associated With Facial Nerve Dysfunction; Facial Asymmetry; Synkinesis
Keywords: Facial paralysis; Facial synkinesis; Botulinum toxin
MeSH Terms: conditions — Facial Nerve Injuries; Facial Asymmetry; Synkinesis; Facial Paralysis | interventions — Botulinum Toxins, Type A; abobotulinumtoxinA; incobotulinumtoxinA

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- OnabotulinumtoxinA Injectable Product (Active Comparator): onabotulinumtoxinA (Botox®, Allergan) administered for n=15 total treatments. Each patient in this arm was administered the Synkinesis Assessment Questionnaire (SAQ) to assess severity of synkinesis pre-treatment. SAQ was administered again at 1, 2, and 4 weeks post-treatment and improvements were compared to the other arms of the study.
  Interventions: Drug: OnabotulinumtoxinA Injectable Product
- AbobotulinumtoxinA Injectable Product (Active Comparator): abobotulinumtoxinA (Dysport®, Medicis) administered for n=13 total treatments. Each patient in this arm was administered the Synkinesis Assessment Questionnaire (SAQ) to assess severity of synkinesis pre-treatment. SAQ was administered again at 1, 2, and 4 weeks post-treatment and improvements were compared to the other arms of the study.
  Interventions: Drug: AbobotulinumtoxinA Injectable Product
- Incobotulinumtoxin A Injectable Product (Active Comparator): incobotulinumtoxinA (Xeomin®, Merz) administered for n=10 total treatments. Each patient in this arm was administered the Synkinesis Assessment Questionnaire (SAQ) to assess severity of synkinesis pre-treatment. SAQ was administered again at 1, 2, and 4 weeks post-treatment and improvements were compared to the other arms of the study.
  Interventions: Drug: Incobotulinumtoxin A Injectable Product

INTERVENTIONS:
Drug: OnabotulinumtoxinA Injectable Product — Administered to treat facial synkinesis
  Other Names: Botox
  Arms: OnabotulinumtoxinA Injectable Product
Drug: AbobotulinumtoxinA Injectable Product — Administered to treat facial synkinesis
  Other Names: Dysport
  Arms: AbobotulinumtoxinA Injectable Product
Drug: Incobotulinumtoxin A Injectable Product — Administered to treat facial synkinesis
  Other Names: Xeomin
  Arms: Incobotulinumtoxin A Injectable Product

SUMMARY:
The purpose of this study is to compare the effectiveness of three commercially available botulinum toxin neuromodulators in the treatment of facial synkinesis using patient reported outcome measures.

DETAILED DESCRIPTION:
Quality assurance:

Data is entered in to a spreadsheet as it is extracted exactly from the electronic medical record. During review of the findings, the data is again checked against the medical record to ensure accuracy. Botulinum toxin types are also verified with scanned copies of the botulinum toxin injection sheet which is filled out and scanned in to the medical record at the time of treatment.

Data dictionary:

Not necessary as limited new terminology is used and all understood among the research group. Additional terminology is clearly described for the trial participants and described in the manuscript reporting the results of the study.

Recruitment:

Patients with facial synkinesis who were appropriate candidates for botulinum toxin chemodenervation therapy were offered voluntary participation in this trial. Patients who had returned to their baseline SAQ score after a minimum of 12 weeks since their previous treatment were permitted to re-enroll in the study for subsequent treatments.

Data collection:

At 1, 2, and 4 weeks post treatment, patients were again administered the SAQ. SAQ scores were calculated for each follow up time point. The average SAQ score in each treatment group (onabotulinumtoxinA, abobotulinumtoxinA, and incobotulinumtoxinA) for each week was calculated, as well as the average improvement in SAQ scores.

Data management:

Data were initially recorded and stored in the secure, password protected, electronic medical record. Data were then extracted from the electronic medical record to a secure Excel spreadsheet stored on a password protected computer. Only the principal investigator and those researchers involved in data analysis and interpretation were provided access to this data. Names and identifiable information were excluded from this spreadsheet so that the information could not be linked back to specific patients.

Data analysis:

Data were analyzed by first organizing the data in Excel, within the original spreadsheet used to record data, then exporting this data in to Prism 6 for Windows (GraphPad Software). Using Prism 6, characteristics of the data were assessed and statistical calculations were performed to determine significance of comparisons between groups. Details of these statistical tests are described below.

Reporting for adverse events:

Adverse events were recorded in the electronic medical record at each follow-up visit. These were then noted in the data spreadsheet as well to keep track of any events that had occurred over the study period. Minor adverse effects reported during the study included redness, bruising, swelling, and fullness at the injection sites which were not felt to be significant or noted to be qualitatively different between products. No major adverse treatment effects were reported during the course of the study.

Change management:

There were no significant changes to study protocol over the course of the study.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect:

https://www.dssresearch.com/knowledgecenter/toolkitcalculators/statisticalpowercalculators.aspx At an alpha level of 0.05, an estimated standard deviation of 10, an estimated average of SAQ 44 and comparison/test value of SAQ 55, a sample size was calculated of approximately 400. We were unable to obtain this sample size after nearly 3 years of enrolment from July 2012 to March 2015. However, despite not reaching this estimated sample size, we did identify a statistically significant finding at alpha level of 0.05 and with a standard deviation of approximately 10-15 per group.

Plan for missing data to address situations where variables are reported as missing, unavailable, "non-reported," uninterpretable, or considered missing because of data inconsistency or out-of-range results:

Patients without follow-up at the post-treatment time points of 1, 2, and 4 weeks were excluded and therefore no missing data was expected for SAQ values. The plan for any missing data in the study was to leave the data point as missing without attempts to imputate the value or otherwise correct for missingness.

Statistical analysis plan describing the analytical principles and statistical techniques to be employed in order to address the primary and secondary objectives, as specified in the study protocol or plan:

The average SAQ score in each treatment group (onabotulinumtoxinA, abobotulinumtoxinA, and incobotulinumtoxinA) for each week was calculated, as well as the average improvement in SAQ scores. Lower SAQ scores represented less severe patient reported disease. Percent improvement in SAQ score was calculated for each time point as the average post-treatment score divided by the average pre-treatment score for the treatment group, subtracted from 1. The SAQ scores for each time point and treatment groups were found to be normally distributed (passing both the D'Agostino & Pearson omnibus normality test as well as Shapiro-Wilk normality test) allowing for an assumption of Gaussian distribution in our following tests of statistical significance. Comparisons between treatments, and between time points within treatment groups were made with a one-way ANOVA followed by appropriate follow-up test for multiple comparisons. Comparisons within treatment groups between each follow-up time point, and the control pre-treatment time point were made using the Dunnett test (compares every mean to a control mean), whereas comparisons of different treatments at a given time point were made with the Tukey test (compares every mean to every other mean). A threshold of p ≤ 0.05 was used for statistical significance.

Patients who had returned to their baseline SAQ score after a minimum of 12 weeks since their previous treatment were permitted to re-enroll in the study for subsequent treatments. Twenty-seven patients were studied, and 6 of these 27 were enrolled multiple times accounting for 11 of the 38 treatments studied. To ensure the baseline SAQ scores of these patients receiving repeat treatments did not differ from patients receiving a single treatment, the average pre-treatment SAQ score for patients undergoing repeat treatments was compared to the average pre-treatment SAQ score of single treatment patients for each type of botulinum toxin neuromodulator. These groups were evaluated for normality of distribution by the same method as described above, with single treatment patients passing tests of normality; normality for the repeat patients could not be determined due to the small number of treatments for each of these patients. Statistical comparisons were then made between the pre-treatment SAQ scores for repeat treatment patients and the respective (same type of botulinum toxin) single treatment patients. In order to preference type I error and identify any possible difference between these groups, we made an assumption of normality and used a one-way ANOVA followed by a Holm-Sidak multiple comparison test. The Holm-Sidak method was chosen as it has more power to identify significant differences than other possible methods such as that of Bonferroni.

ELIGIBILITY:
Inclusion Criteria:

* Facial synkinesis

Exclusion Criteria:

* Previous complication from botulinum toxin neuromodulator injection
* Inability to understand or complete the SAQ survey
* Inability to participate in follow-up
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Preston D Ward, MD, Principal Investigator — University of Utah

IPD SHARING:
Plan to Share IPD: Yes
IPD is to be shared among the first author of the study and the principal investigator for purposes of data acquisition and analysis. This data will be limited to that necessary to addressing the research question, specifically, the type of botulinum toxin used for treatment, the dates of treatment, and the SAQ scores at the pre-treatment, and post-treatment follow-up visits. Any adverse events related to treatment will also be available.

REFERENCES:
- [Background] Choi KH, Rho SH, Lee JM, Jeon JH, Park SY, Kim J. Botulinum toxin injection of both sides of the face to treat post-paralytic facial synkinesis. J Plast Reconstr Aesthet Surg. 2013 Aug;66(8):1058-63. doi: 10.1016/j.bjps.2013.04.012. Epub 2013 May 15. PMID 23683725
- [Background] Nettar KD, Yu KC, Bapna S, Boscardin J, Maas CS. An internally controlled, double-blind comparison of the efficacy of onabotulinumtoxinA and abobotulinumtoxinA. Arch Facial Plast Surg. 2011 Nov-Dec;13(6):380-6. doi: 10.1001/archfacial.2011.37. Epub 2011 Jun 20. PMID 21690460
- [Background] Saad J, Gourdeau A. A direct comparison of onabotulinumtoxina (Botox) and IncobotulinumtoxinA (Xeomin) in the treatment of benign essential blepharospasm: a split-face technique. J Neuroophthalmol. 2014 Sep;34(3):233-6. doi: 10.1097/WNO.0000000000000110. PMID 24739994
- [Background] Mehta RP, WernickRobinson M, Hadlock TA. Validation of the Synkinesis Assessment Questionnaire. Laryngoscope. 2007 May;117(5):923-6. doi: 10.1097/MLG.0b013e3180412460. PMID 17473697
- [Background] Filipo R, Spahiu I, Covelli E, Nicastri M, Bertoli GA. Botulinum toxin in the treatment of facial synkinesis and hyperkinesis. Laryngoscope. 2012 Feb;122(2):266-70. doi: 10.1002/lary.22404. Epub 2012 Jan 17. PMID 22252570
- [Background] Armstrong MW, Mountain RE, Murray JA. Treatment of facial synkinesis and facial asymmetry with botulinum toxin type A following facial nerve palsy. Clin Otolaryngol Allied Sci. 1996 Feb;21(1):15-20. doi: 10.1111/j.1365-2273.1996.tb01018.x. PMID 8674216
- [Background] Naumann M, Albanese A, Heinen F, Molenaers G, Relja M. Safety and efficacy of botulinum toxin type A following long-term use. Eur J Neurol. 2006 Dec;13 Suppl 4:35-40. doi: 10.1111/j.1468-1331.2006.01652.x. PMID 17112348
- [Derived] Thomas AJ, Larson MO, Braden S, Cannon RB, Ward PD. Effect of 3 Commercially Available Botulinum Toxin Neuromodulators on Facial Synkinesis: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2018 Mar 1;20(2):141-147. doi: 10.1001/jamafacial.2017.1393. PMID 28973094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were prospectively enrolled from July 2012 to March 2015. All patients 18 years and older with facial synkinesis, who presented to our tertiary care Facial Nerve Center for treatment and were appropriate candidates for botulinum toxin chemodenervation therapy, were offered voluntary participation.
Pre-assignment Details: Exclusion criteria included previous complication from botulinum toxin neuromodulator injection, inability to understand or complete the SAQ survey, inability to participate in follow-up, and pregnancy. Informed consent was obtained from each patient before enrollment in the study.
Period: Overall Study
Arm/Group | OnabotulinumtoxinA Injectable Product | AbobotulinumtoxinA Injectable Product | Incobotulinumtoxin A Injectable Product
Started | 28 | 21 | 22
Completed | 15 | 13 | 10
Not Completed | 13 | 8 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OnabotulinumtoxinA Injectable Product | AbobotulinumtoxinA Injectable Product | Incobotulinumtoxin A Injectable Product | Total
Number analyzed (Participants) | 15 | 13 | 10 | 38
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [24 to 76] | 52.1 [21 to 83] | 53.2 [32 to 73] | 49.1 [21 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 6 | 23
  Male | 5 | 6 | 4 | 15
Pre-treatment SAQ score [Mean (Standard Deviation); unit: units on a scale] — The Synkinesis Assessment Questionnaire (SAQ) was used to assess severity of facial synkinesis in this study. SAQ scores are calculated as the sum of scores for 9 questions, which each is scored from 1 to 5, divided by 45 and multiplied by 100. The total score therefore can range from 20 to 100. Lower SAQ scores represent less severe facial synkinesis, and higher scores more severe. We report here the mean total SAQ score each group. For additional information on the SAQ for facial synkinesis see Mehta et al. published in Laryngoscope in May 2007 (PMID: 17473697).
  units on a scale | 79.6 (15.1) | 70.1 (15.3) | 69.6 (9.7) | 73.7 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Synkinesis Assessment Questionnaire (SAQ) Scores
Description: The previously validated instrument, Synkinesis Assessment Questionnaire (SAQ), was administered in order to evaluate patient-perceived severity of synkinesis. This instrument was used for each of the three treatment arms and change in scores from baseline were compared at each time point between arms.
  SAQ scores are calculated as the sum of scores for 9 questions, which each is scored from 1 to 5, divided by 45 and multiplied by 100. The total score therefore can range from 20 to 100. Lower SAQ scores represent less severe facial synkinesis, and higher scores more severe. We report here the mean total SAQ score each group. For additional information on the SAQ for facial synkinesis see Mehta et al. published in Laryngoscope in May 2007 (PMID: 17473697).
Time Frame: Up to 4 weeks post-treatment. Recorded at pre-treatment, 1 week, 2 weeks, and at 4 weeks.
Population: The Synkinesis Assessment Questionnaire (SAQ) was used to assess severity of facial synkinesis for each group. Total SAQ scores can range from 20 to 100. Lower SAQ scores represent less severe facial synkinesis, and higher scores more severe.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OnabotulinumtoxinA Injectable Product | AbobotulinumtoxinA Injectable Product | Incobotulinumtoxin A Injectable Product
Number analyzed (Participants) | 15 | 13 | 10
units on a scale
  1 week post-treatment SAQ score | 45.9 (13.9) | 38.8 (10.8) | 51.3 (12.6)
  2 weeks post-treatment SAQ score | 45.2 (15.4) | 37.6 (12.2) | 49.8 (11.8)
  4 weeks post-treatment SAQ score | 46.4 (15.4) | 40.3 (16.0) | 58.0 (11.6)

2. Secondary Outcome: Adverse Events
Description: We hypothesized that common minor events such as bruising and swelling at injection sites would occur equally for all treatment arms, but that no major adverse treatment effects would occur for any of the treatment arms. Major events are recorded here.
Time Frame: Up to 4 weeks post-treatment. Recorded at pre-treatment, 1 week, 2 weeks, and at 4 weeks.
Measure: Number; unit: Adverse Events
Arm/Group | OnabotulinumtoxinA Injectable Product | AbobotulinumtoxinA Injectable Product | Incobotulinumtoxin A Injectable Product
Number analyzed (Participants) | 15 | 13 | 10
Adverse Events | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | OnabotulinumtoxinA Injectable Product | AbobotulinumtoxinA Injectable Product | Incobotulinumtoxin A Injectable Product
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 0/15 | 0/13 | 0/10

LIMITATIONS AND CAVEATS:
Re-enrollment of patients already treated with botulinum toxin for synkinesis (treated as unique patients); small sample size of patients/treatments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No